CLINICAL TRIAL: NCT04675827
Title: De-Escalation of Adjuvant Chemotherapy in HER2-positive, Estrogen Receptor-negative, Node-negative Early Breast Cancer Patients Who Achieved Pathological Complete Response After Neoadjuvant Chemotherapy and Dual HER2 Blockade
Brief Title: De-escalation Adjuvant Chemo in HER2+/ER-/node-neg Early BC Patients Who Achieved PCR After Neoadjuvant Chemo & Dual HER2 Blockade
Acronym: Decrescendo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Serious concerns on the slow recruitment of the study that impacts the robustness of the scientific rationale and the study financial provision. It aims to assess carefully the situation and to evaluate the potential solutions to overcome the issues.
Sponsor: Jules Bordet Institute (Other)
Collaborators: Breast International Group (Other); Hoffmann-La Roche (Industry); International Drug Development Institute (Other); Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IJB-EBC-Decrescendo-2020
Record Dates: First submitted 2020-11-25; First posted 2020-12-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive Breast Cancer; ER-Negative Breast Cancer; PR-Negative Breast Cancer; Node-negative Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Injections, Subcutaneous; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: Eligible subjects will first receive neoadjuvant treatment then surgery. After surgery, subjects who achieve a pCR (RCB score at surgery = 0) will receive adjuvant pertuzumab and trastuzumab FDC SC for additional 14 cycles. Those with residual invasive disease (RCB score at surgery ≥ 1) will receive salvage adjuvant T-DM1 for 14 cycles. In subjects with RCB score as ≥2, 3 to 4 cycles of anthracycline-based chemotherapy may be administered, at the investigator's discretion, before the administration of T-DM1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RCB = 0 (Experimental): Treatment administration: adjuvant pertuzumab + trastuzumab (P+T) fixed dose combination (FDC) SC for 14 cycles.
  Sub-study: 121 of the subjects who achieved a pCR (thus assigned to continue treatment with P+T FDC SC) will be randomised at a 1:1 ratio to receive 3 cycles of P+T FDC SC in the hospital, followed by 3 cycles in another setting outside the hospital, or to the same treatment starting with 3 cycles outside the hospital followed by 3 cycles in the hospital (treatment cross-over period). After the first 6 cycles of adjuvant treatment, subjects will be asked to choose between continuing treatment (for the remaining 8 cycles, for a total of 14 cycles) within or outside the hospital, according to their preference (treatment continuation period). Subjects can request to change from outside the hospital to in the hospital administration (and vice-versa) at any moment during the treatment continuation period, but not in the treatment cross-over period.
  Interventions: Drug: Pertuzumab and tratuzumab fixed dose combination
- RCB > 0 (Experimental): Treatment administration:adjuvant T-DM1 for 14 cycles. In subjects whose residual invasive disease is classified per Residual Cancer Burden (RCB) score as ≥2, 3 to 4 cycles of anthracycline-based chemotherapy may be administered, at the investigator's discretion, before the 14 cycles of T-DM1.
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Pertuzumab and tratuzumab fixed dose combination — Treatment administration: adjuvant pertuzumab and trastuzumab fixed dose combination SC for 14 cycles
  Other Names: Adjuvant pertuzumab + trastuzumab FDC SC for 14 cycles; Fixed-dose combination of Perjeta and Herceptin for subcutaneous injection for 14 cycles
  Arms: RCB = 0
Drug: Trastuzumab emtansine — Treatment administration: adjuvant T-DM1 for 14 cycles.
  Other Names: Adjuvant T-DM1
  Arms: RCB > 0

SUMMARY:
DECRESCENDO is a multicentre, open-label, dual-phase single-arm phase II de-escalation study evaluating neoadjuvant treatment with 12 administrations of weekly IV paclitaxel 80 mg/m2 (or IV docetaxel 75 mg/m2 every 3 weeks for 4 cycles) combined with subcutaneous (SC) fixed dose combination (FDC) of pertuzumab and trastuzumab (loading dose of 1200 mg pertuzumab and 600 mg trastuzumab, followed by 600 mg pertuzumab and 600 mg trastuzumab) every 3 weeks for 4 cycles.

Surgery will be performed according to local guidelines in all subjects after neoadjuvant treatment.

After surgery, subjects who achieve a pCR (defined as pT0/Tis pN0) will receive adjuvant pertuzumab and trastuzumab FDC SC for additional 14 cycles. Subjects with residual invasive disease will receive salvage adjuvant trastuzumab emtansine (T-DM1, 3.6 mg/kg, IV every 3 weeks) for 14 cycles. In subjects whose residual invasive disease is classified per RCB score as ≥2, 3 to 4 cycles of anthracycline-based chemotherapy may be administered, at the investigator's discretion, before the 14 cycles of T-DM1.

If histopathological analysis finds that the surgical specimen from a subject with residual disease is ER-positive and/or PR-positive, adjuvant endocrine therapy may be administered concomitantly with study treatment, at the investigator's discretion and according to local guidelines.

Adjuvant radiotherapy will be mandatory after breast-conserving surgery, whereas it will be performed according to local guidelines after mastectomy, and it will be administered concomitantly with pertuzumab and trastuzumab FDC SC in subjects who achieve a pCR, and concomitantly with T-DM1 in subjects with residual invasive disease (after anthracycline-based chemotherapy in subjects assigned to receive this treatment).

DETAILED DESCRIPTION:
DECRESCENDO is a multicentre, open-label, dual-phase single-arm phase II de-escalation study evaluating neoadjuvant treatment with 12 administrations of weekly intravenous (IV) paclitaxel 80 mg/m2 (or IV docetaxel 75 mg/m2 every 3 weeks for 4 cycles) combined with subcutaneous (SC) fixed dose combination (FDC) of pertuzumab and trastuzumab (loading dose of 1200 mg pertuzumab and 600 mg trastuzumab, followed by 600 mg pertuzumab and 600 mg trastuzumab) every 3 weeks for 4 cycles.

Surgery will be performed according to local guidelines in all subjects after neoadjuvant treatment.

After surgery, subjects who achieve a pathologic complete response (pCR, defined as pT0/Tis pN0) will receive adjuvant pertuzumab and trastuzumab FDC SC for additional 14 cycles. Subjects with residual invasive disease will receive salvage adjuvant trastuzumab emtansine (T-DM1, 3.6 mg/kg, IV every 3 weeks) for 14 cycles. In subjects whose residual invasive disease is classified per Residual Cancer Burden (RCB) score as ≥2, 3 to 4 cycles of anthracycline-based chemotherapy may be administered, at the investigator's discretion, before the 14 cycles of T-DM1.

If histopathological analysis finds that the surgical specimen from a subject with residual disease is ER-positive and/or PR-positive, adjuvant endocrine therapy may be administered concomitantly with study treatment, at the investigator's discretion and according to local guidelines.

Adjuvant radiotherapy will be mandatory after breast-conserving surgery, whereas it will be performed according to local guidelines after mastectomy, and it will be administered concomitantly with pertuzumab and trastuzumab FDC SC in subjects who achieve a pCR, and concomitantly with T-DM1 in subjects with residual invasive disease (after anthracycline-based chemotherapy in subjects assigned to receive this treatment).

Patients' tumour intrinsic subtype will be determined based on analysis of the PAM50 gene signature. The PAM50 gene signature, which measures the expression of 50 genes to classify tumours into 1 of 4 intrinsic subtypes (luminal A, luminal B, HER2-enriched, and basal-like), will be assessed in formalin-fixed paraffin embedded (FFPE) samples obtained at baseline. While a tumour biopsy sample must be available prior to enrolment, the PAM50 results will be generated centrally post enrolment and subsequently used to assess the primary endpoint of the study, which is the 3-year recurrence-free survival (RFS) rate in the subpopulation of subjects with HER2-enriched tumours who achieve a pCR after the neoadjuvant phase of the study.

Sub-study:

The flexible care sub-study is an open-label, randomised phase II study to be conducted in selected sites from some of the countries that participate in DECRESCENDO. After completion of neoadjuvant treatment and surgery in the main study, 121 of the subjects who achieved a pCR and thus are assigned to continue treatment with pertuzumab and trastuzumab FDC SC will be randomised at a 1:1 ratio to receive 3 cycles of pertuzumab and trastuzumab FDC SC every 3 weeks in the hospital, followed by 3 cycles in another setting outside the hospital, or to the same treatment starting with 3 cycles outside the hospital followed by 3 cycles in the hospital (treatment cross-over period). After the first 6 cycles of adjuvant treatment, subjects will be asked to choose between continuing treatment (for the remaining 8 cycles, for a total of 14 cycles) within or outside the hospital, according to their preference (treatment continuation period). Subjects can request to change from outside the hospital to in the hospital administration (and vice-versa) at any moment during the treatment continuation period, but not in the treatment cross-over period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age ≥18 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
4. Subjects whose tumour measures ≥15 mm and ≤50 mm, according to clinical staging performed with imaging exams (either mammography, ultrasound or breast magnetic resonance imaging [MRI]).
5. Must have histologically confirmed diagnosis of HER2-positive and ER-negative/PR-negative breast cancer (analysis performed by the local laboratory).

   1. HER2-positive defined as a score of 3+ in IHC or a positive ISH (ratio of HER2 copy number/chromosome 17 ≥2 or average HER2 copy number ≥6 signals per cell).
   2. ER-negative/PR-negative defined as estrogen receptor and progesterone receptor nuclear staining <1% by IHC.

   Note: patients with micro-invasive carcinoma or ductal carcinoma in situ (DCIS) without invasive disease are not eligible.
6. Subjects with multifocal or multicentric invasive disease are eligible as long as all the biopsiable lesions can be characterised and are confirmed to be HER2-positive and ER and PR negative.

   Note: In the case of multifocal or multicentric disease, only the biopsy from the largest lesion should be provided.
7. Node-negative disease (N0): no axillary lymph nodes identifiable at ultrasound, or in case of suspect axillary lymph nodes are identified, fine-needle aspiration or core biopsy must be carried out to confirm that axillary status is negative. Axillary micrometastases (i.e., if the greatest diameter of the nodal metastasis in a sentinel node is 0.2 mm or less) are not allowed.
8. Serum pregnancy test (for women of childbearing potential) negative within 7 days prior to treatment start.
9. Women of childbearing potential must agree to use 1 highly effective non-hormonal contraceptive method with a failure rate of less than 1% per year from the signing of the ICF until at least 7 months after last dose of study drugs; or they must totally abstain from any form of sexual intercourse. Men with a partner of childbearing potential must agree to use condom in combination with a spermicidal foam, gel, film, cream, or suppository, and agreement to refrain from donating sperm, during the course of this study and for at least 7 months after the last administration of study treatment.
10. Adequate bone marrow and coagulation functions as defined below:

    * Absolute neutrophil count ≥1500 /µL or 1.5x109/L
    * Haemoglobin ≥9 g/dL (blood transfusions to reach these levels of haemoglobin are allowed)
    * Platelets ≥100,000/µL or 100x109/L
    * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 ×ULN
11. Adequate liver function as defined below:

    * Serum total bilirubin ≤1.5 x ULN. In case of known Gilbert's syndrome ≤3xUNL is allowed
    * AST (SGOT) and ALT (SGPT) ≤2.5 x ULN
    * Alkaline phosphatase ≤2.5 x ULN
12. Adequate renal function as defined below:

    • Creatinine ≤1.5 x UNL or creatinine clearance >60 mL/min/1.73 m2
13. Completion of all necessary screening procedures within 28 days prior to enrolment.
14. Adequate cardiac function, defined as a left ventricular ejection fraction ≥55% estimated by echocardiogram (ECHO) or multiple-gated acquisition scintigraphy (MUGA).
15. Availability of a pre-treatment tumour biopsy sample as specified below:

    * At least one FFPE tumour block must be available for central evaluation. Whenever possible, two FFPE tumour blocks should be available (preferred).
    * If a block cannot be provided, 25 unstained FFPE slides of 4 µm thickness from the pre-treatment tumour biopsy must be provided as an alternative. These slides must be freshly cut prior the shipment to the sponsor.
    * In either case, the local pathologist must evaluate an H&E stained slide to ensure that the tumour surface is at least 4 mm² and that tumour cellularity is ≥10%.

    Note 1: Tumour biopsy must be sent to the central research laboratory as soon as the patient is confirmed by the local investigator to be eligible for the study.

    Note 2: the inclusion of the subject is only based on local assessments. A central review of HER2, ER, and PR status will be performed at posteriori for quality control purposes.
16. Signed Informed Consent form (ICF) obtained prior to any study related procedure.
17. Subject is willing and able to comply with the protocol for the duration of the study including treatment and scheduled visits and examinations.

    Inclusion criterion applicable to FRANCE only:
18. Affiliated to the French Social Security System.

Exclusion Criteria:

1. Pregnant and/or lactating women.
2. Bilateral invasive breast cancer.
3. Evidence of metastatic breast cancer: all subjects must have had a CT/MRI scan of the thorax/abdomen/pelvis to rule out metastatic breast cancer prior to enrolment. FDG/PET-CT can be used as an alternative to replace all the exams above. A screening bone scan must have been done if ALP and/or corrected calcium levels were above the institutional upper limits at screening (if PET/CT was used as an alternative imaging exam, a bone scan and/or CT/MRI is not required).
4. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the investigator's opinion, may interfere with completion of the study.
5. Previous exposure to any anti-HER2 treatment.
6. Concomitant exposure to any investigational products as part of a clinical trial within 30 days prior to enrolment.
7. Subject with second primary malignancies diagnosed ≤ 5 years before enrolment in the study. Exceptions are: adequately treated non-melanoma skin cancer, in situ cancer of the cervix, ductal carcinoma in situ of the breast, and any other solid or haematological tumour diagnosed > 5 years before enrolment and for which no chemotherapy and no systemic treatment were necessary, with no evidence of disease recurrence.
8. Resting electrocardiogram (ECG) with QTc >470 msec detected on at 2 or more time points within a 24-hour period, or family history of long QT syndrome.
9. Serious cardiac illness or medical conditions including, but not confined to, the following:

   * History of NCI CTCAE (v4) Grade ≥ 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) Class ≥ II
   * High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate = or > 100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block, such as second degree AV-block Type 2 [Mobitz 2] or third-degree AV-block) - Serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality
   * Angina pectoris requiring anti-anginal medication
   * Clinically significant valvular heart disease
   * Evidence of transmural infarction on ECG
   * Evidence of myocardial infarction within 12 months prior to randomization
   * Poorly controlled hypertension (i.e., systolic > 180 mm Hg or diastolic > 100 mmHg)
10. History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe LVSD, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome.
11. Peripheral neuropathy (CTCAE version 5) grade ≥2.
12. Major surgery within 14 days prior to enrolment.
13. Subject with HIV, Hepatitis B or Hepatitis C infection documented by serology, except for those subjects with a previous exposure to Hepatitis B who developed an effective immune response (HBSAg-negative and anti-HBS-positive).
14. Previous allogeneic bone marrow transplant.
15. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAE grade ≥3).
16. Subjects who received live attenuated vaccines within 14 days before enrolment.

    Exclusion criterion applicable to FRANCE only:
17. Vulnerable persons according to the article L.1121-6 of the CSP, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the CSP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
3-year RFS in HER2-enriched subjects who achieve a pCR | 3 years
  3-year RFS, defined as the time from enrolment until the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence, death from breast cancer, death attributable to any cause other than breast cancer, death from unknown cause; in subjects with HER2-enriched, ER-negative/PR-negative, clinically node-negative breast cancers who achieve a pCR after neoadjuvant treatment.

SECONDARY OUTCOMES:
3-year RFS in all subjects who achieve a pCR. | 3 years
  3-year RFS in all subjects who achieve a pCR.
5-year RFS in all subjects who achieve a pCR. | 5 years
  5-year RFS in all subjects who achieve a pCR.
pCR (in the overall population) | during procedure
  To assess pCR rates in the overall population and by primary tumour dimension. pCR (in the overall population) is defined as the absence of residual invasive tumour in the breast and axillary lymph nodes (pT0/Tis pN0) at surgery as per the local anatomo-pathological report.
3-year RFS (survival rates) | 3 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 3-year RFS The RFS is defined as the time from enrolment until the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence, death from breast cancer, death attributable to any cause other than breast cancer, death from unknown cause
3-year invasive disease-free survival (iDFS) (survival rates) | 3 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 3-year invasive disease-free survival (iDFS) The iDFS is defined as the time from enrolment until the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence, death from breast cancer, death attributable to any cause other than breast cancer, death from unknown cause, invasive contralateral breast cancer, second primary invasive cancer (non-breast)
3-year distant disease-free survival (dDFS) (survival rates) | 3 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  urvival rates: - 3-year distant disease-free survival (dDFS) The dDFS defined as the time from enrolment until the first occurrence of one of the following events: distant recurrence; death from breast cancer; death from non-breast cancer cause; death from unknown cause; second primary invasive cancer (non-breast);
3-year overall survival (OS) (survival rates) | 3 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 3-year overall survival (OS) The OS defined as the time from enrolment until the first occurrence of one of the following events: death from breast cancer, death from non-breast cancer cause, death from unknown cause
Recurrence-free interval (RFI) (Time) | 3 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Time: Recurrence-free interval (RFI) The RFI is defined as the time interval between enrolment and the occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence; death from breast cancer
5-year RFS (survival rates) | 5 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 5-year RFS The RFS is defined as the time from enrolment until the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence, death from breast cancer, death attributable to any cause other than breast cancer, death from unknown cause
5-year invasive disease-free survival (iDFS) (survival rates) | 5 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 5-year invasive disease-free survival (iDFS) The iDFS is defined as the time from enrolment until the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence, death from breast cancer, death attributable to any cause other than breast cancer, death from unknown cause, invasive contralateral breast cancer, second primary invasive cancer (non-breast)
5-year distant disease-free survival (dDFS) (survival rates) | 5 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 5-year distant disease-free survival (dDFS) The dDFS defined as the time from enrolment until the first occurrence of one of the following events: distant recurrence; death from breast cancer; death from non-breast cancer cause; death from unknown cause; second primary invasive cancer (non-breast);
5-year overall survival (OS)(survival rates) | 5 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Survival rates: - 5-year overall survival (OS) The OS defined as the time from enrolment until the first occurrence of one of the following events: death from breast cancer, death from non-breast cancer cause, death from unknown cause
Recurrence-free interval (RFI) (time) | 5 years
  In all population, the sub-group analysis according to the pathological response (pCR versus residual disease) and stratified by tumour size (T1 versus T2) for following outcomes:
  Time: Recurrence-free interval (RFI) The RFS is defined as the time from enrolment until the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence, local/regional invasive recurrence, distant recurrence, death from breast cancer, death attributable to any cause other than breast cancer, death from unknown cause
Number of participants experiencing an Adverse Event | study treatment plus follow-up of 30 days ( Time Frame: Up to approximately 17 months )
  An adverse event (AE) is any untoward medical occurrence in a subject or clinical investigation subject receiving/undergoing the study treatments (paclitaxel (or docetaxel), pertuzumab and trastuzumab FDC SC, T-DM1, surgery, radiotherapy) and which does not necessarily have a causal relationship with these study treatments. The number of participants who experience an AE (including 1 month of safety follow up) will be presented. The intensity of all AEs will be graded according to the CTCAE version 5 on a five-point scale (Grade 1 to 5).
Number of participants experiencing an Serious Adverse Event | through study completion estimated 60 months
  A serious adverse event (SAE) is any untoward medical occurrence that results in any of the following outcomes: Death; Life-threatening; Subject hospitalisation or prolongation of existing hospitalisation; Persistent or significant disability/incapacity; Congenital anomaly/birth defect. The number of participants who experience any SAE while receiving paclitaxel (or docetaxel), pertuzumab and trastuzumab FDC SC, T-DM1, surgery, radiotherapy (including 1 months of safety follow up) with or without the relationship to IMPs will be presented. During survival follow-up, only SAE related to IMPs will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Piccart, PD, PhD, Study Chair — Jules Bordet Institute
Locations (85):
- Australia (23):
  - Icon Cancer Centre Wesley, Auchenflower
  - Ballarat Health Services, Ballarat
  - Bendigo Hospital, Bendigo
  - Sunshine Coast University Hospital, Birtinya
  - Box Hill Hospital, Box Hill
  - Chris O'Brien Lifehouse, Camperdown
  - Monash Medical Centre (Clayton), Clayton
  - Coffs Harbour Health Campus, Coffs Harbour
  - Concord Repatriation General Hospital, Concord
  - Townsville University Hospital, Douglas
  - Lake Macquarie Private Hospital, Gateshead
  - Gosford Hospital, Gosford
  - Royal Brisbane and Women's Hospital, Herston
  - Icon Cancer Centre Hobart, Hobart
  - Liverpool Hospital, Liverpool
  - Peter MacCallum Cancer Centre, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Macquarie University, North Ryde
  - Mater Hospital, North Sydney
  - Sunshine Hospital, Saint Albans
  - Calvary Mater Newcastle, Waratah
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (8):
  - GZA Ziekenhuisen Campus Sint-Augustinus - Iridium Kankernetwerk, Antwerp, Wilrijk
  - OLV ziekenhuis, Aalst
  - Cliniques Universtaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Heilig Hartziekenhuis, Lier
  - Centre Hospitalier Chretien MontLegia, Liège
  - CHU UCL Namur Sainte-Elisabeth, Namur
- France (31):
  - Institut de Cancérologie de l'Ouest - Angers, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU Morvan, Brest
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Hopital Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - GHBS Lorient, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH Annecy Genevois, Metz-Tessy
  - Centre de Cancerologie du Grand Montpellier, Montpellier
  - Hopital privé du Confluent, Nantes
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Hopital Tenon, Paris
  - Institut Curie - Paris, Paris
  - CH Perpignan, Perpignan
  - Hopital Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Institut Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Saint-Cloud, Saint-Cloud
  - Clinique Saint Anne, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Sheba Medical Center, Ramat Gan, Israel
- South Korea (16):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - CHA bundang Medical Center, Seongnam-si
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea university anam hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul ST. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Switzerland (6):
  - Hirslanden Klinik - Tumor Zentrum, Aarau
  - Kantonsspital Baden, Baden
  - Universitatsspital Basel, Basel
  - Kantonsspital Frauenfeld/Frauenklinik, Frauenfeld
  - Hopital Daler - Centre du Sein, Fribourg
  - Kantonsspital Winterthur, Winterthur